CLINICAL TRIAL: NCT00006072
Title: A Study of Rituxan in the Treatment of Polyneuropathies Associated With Serum IgM Autoantibodies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Genentech, Inc. (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: NCRR-M01RR00036-0690; M01RR000036 (NIH)
Record Dates: First submitted 2000-07-25; First posted 2000-07-26 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-07

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Rituximab

INTERVENTIONS:
Drug: Rituxan

SUMMARY:
Peripheral neuropathies cause weakness and sensory loss that can produce severe disability. Some neuropathies are immune-mediated and associated with antibodies. It has been postulated that Rituxan treatment may reduce the level of antibody production limiting the loss of muscle strength and hence improve activities of daily living. The purpose of this open-label study (all participants get Rituxan and not placebo) is to determine the safety and effectiveness of Rituxan in the treatment of polyneuropathies associated with serum IgM autoantibodies in those who have already been treated with one course of Rituxan. Subjects will be treated on the in-patient Clinical Research Center with Rituxan for two treatments one week a part and then individual treatments every 10 weeks for one year. The effectiveness of Rituxan will be followed by looking for increases in muscle strength and decreases in the serum IgM autoantibodies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of characteristic peripheral neuropathy by appropriate history, physical examination, nerve conduction findings and serum autoantibodies.
* Serum anti-GM1 on anti-MAG antibodies present at high titers in serum, continued by testing in the neuromuscular clinical laboratory at Washington University.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult